CLINICAL TRIAL: NCT06045988
Title: Automated, Assistive, Non-Contact Sleep Quality Monitor for Individuals With Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Innovative Design Labs (Industry); University of Minnesota (Other); Mayo Clinic (Other); National Institute on Aging (NIA) (NIH); Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Kathleen T. Unroe, Professor of Medicine, Geriatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15771; 2R44AG058339-02A1 (NIH)
Record Dates: First submitted 2023-08-07; First posted 2023-09-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Dementia; Sleep Disturbance
Keywords: Sleep Assessment; Sleep Disorder; Technology; Dementia; Long-Term Care; Sleep Monitoring
MeSH Terms: conditions — Alzheimer Disease; Dementia; Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Long-Term Care Facility Residents with Alzheimer's Disease or other Related Dementias (Experimental)
  Interventions: Device: Non-Contact Sleep Quality Monitor System

INTERVENTIONS:
Device: Non-Contact Sleep Quality Monitor System — Residents of long-term care facilities with Alzheimer's or other related dementias will utilize a sleep monitoring device for the four-week period they are involved in the study.

SUMMARY:
This study seeks to evaluate the utility and efficacy of the Non-Contact Sleep Quality Monitor System when used to monitor the sleep quality of individuals living in long-term care (LTC) with either Alzheimer's Disease (AD) or Alzheimer's Disease Related Dementia (ADRD). This before-after comparison trial will be conducted in several LTC facilities to evaluate the effect access to System Sleep Quality Data has on documentation of sleep disorders or treatments and sleep quality change over time for AD/ADRD participants in the intervention group as compared to the control group.

All subjects will undergo sleep quality monitoring for 4-weeks. At the end of the first 2-weeks, research staff and LTC facility staff and medical providers will receive access to sleep monitoring data. We hypothesize that when real-time System Sleep Data is shared with LTC staff or healthcare providers, that sleep disturbances will be more readily detected, leading to timelier, better tailored treatment interventions for sleep disturbances, thereby improving sleep quality and decreasing daytime physical inactivity.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the utility of a Non-Contact Sleep Quality Monitor System and determine the effect that sharing System Sleep Data with long-term care (LTC) staff and healthcare providers has on documentation and treatment of sleep disorders and change in AD/ADRD participant sleep quality. System Sleep Data will be collected for a total of 4-weeks. During the Intervention condition System Sleep Data will be shared for 2-weeks, while in the initial Control condition no System Sleep Data will be shared for 2-weeks. Healthcare providers can prescribe a non-pharmacologic sleep protocol and/or if they so choose, pharmacotherapy to manage sleep disturbances for subjects in either the Intervention or Control condition, in accordance with standard medical practice. The investigators hypothesize that when real-time System Sleep Data is shared with LTC staff or healthcare providers, that sleep disturbances will be more readily detected, leading to timelier, better tailored treatment interventions for sleep disturbances, thereby improving sleep quality and decreasing daytime physical inactivity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's Disease (AD) or Alzheimer's Disease Related Dementias (ADRD)
* Residents of long-term care (LTC) facility study site location for a minimum of 30 days.
* Willingness to consent to study or when a potential participant lacks decision making capacity (determined by LTC facility clinical provider) willingness of a Legally Authorized Representative (LAR) to consent to study participation on potential participant's behalf.

Exclusion Criteria:

* Currently on hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Documentation of sleep disorders or treatment | 4-weeks
  Primary outcome documentation of diagnosis, or evidence of treatment of sleep disorders, will be obtained through review of the medical record. Evidence of such a diagnosis or treatment could be indicated in nursing notes, physician notes, psychoactive or sedative medication changes, new ICD 10 sleep disorder diagnoses, medical orders for sleep studies or sleep medicine consults, all contained in the medical record.

SECONDARY OUTCOMES:
Change in Sleep Quality Over Time: Total Nocturnal Sleep Time (TNST) | 4-weeks
  Total Nocturnal Sleep Time (TNST) will be derived from System Data and Algorithms.
Change in Epworth Sleepiness Scale Total Score Over Time | 4-weeks
  The Epworth Sleepiness Scale is a validated, self-report measure of sleepiness. It is an 8-item questionnaire that measures one's tendency to become sleepy using a scale from 0 (no chance of dozing) to 3 (high chance of dozing). The total score is based on a scale of 0 to 24, with a score of 24 indicating the potential need for medical attention.
Change in QOL-AD Over Time | 4-weeks
  The Quality-Of-Life-Alzheimer's Disease (QOL-AD) instrument is a 13-item questionnaire that measures the domains of physical condition, mood, memory, functional abilities, interpersonal relationships, ability to participate in meaningful activities, financial situation, and global assessments of self as a whole and QOL as a whole.
Attitudes Toward Technology | 4-weeks
  A questionnaire that measures attitudes toward technology created by Jay & Willis 1992.
Technology Acceptance Survey Questionnaire | 4-weeks
  A validated 12-item questionnaire that measures perceptions of technology usefulness and
  usability, derived from Davis 1989
System Usage | 4-weeks
  The total number of days out of 28 that the system collected data, and the number of times the System Sleep Data User Interface was accessed.
Change in Sleep Quality Over Time: Sleep Efficiency (SE) | 4-weeks
  Sleep Efficiency (SE) will be derived from System Data and Algorithms.
Change in Sleep Quality Over Time: Sleep Onset Latency (SOL) | 4-weeks
  Sleep Onset Latency (SOL) will be derived from System Data and Algorithms.
Change in Sleep Quality Over Time: Wake After Sleep Onset (WASO) | 4-weeks
  Wake After Sleep Onset (WASO) will be derived from System Data and Algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Unroe, MD, MHA, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No